CLINICAL TRIAL: NCT01927627
Title: A Phase 2 Study of Enzalutamide in Patients With High-risk Prostate Cancer Who Have Undergone Local Definitive Therapy With Radical Prostatectomy
Brief Title: Enzalutamide in Patients With High-risk Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE12812; NCI-2013-01661 (Other: NCI/CTRP)
Record Dates: First submitted 2013-08-19; First posted 2013-08-22 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Prostate cancer; adenocarcinoma of the prostate; Enzalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enzalutamide (Experimental): Oral therapy with enzalutamide at 160mg (4 capsules) orally once daily (QD).
  Interventions: Drug: enzalutamide

INTERVENTIONS:
Drug: enzalutamide — oral therapy with enzalutamide at 160mg (4 capsules) orally once daily (QD).
  Other Names: XTANDI; MDV3100

SUMMARY:
The purpose of this study is to see how long it takes for prostate cancer to come back in patients who have had surgery to remove their prostate gland (radical prostatectomy), while being treated with enzalutamide (formerly known as MDV3100).

Enzalutamide is known as an androgen-receptor signaling inhibitor, which means that it blocks activity of the male hormone, testosterone. Most prostate cancers are dependent on testosterone for growth. In this study, patients will take enzalutamide after surgery to see if it keeps their cancer from coming back.

DETAILED DESCRIPTION:
This is a pilot phase II study evaluating the clinical activity and safety of Enzalutamide (formerly known as MDV3100) a novel androgen receptor (AR) inhibitor in men with high-risk prostate cancer who have undergone local definitive therapy with radical prostatectomy.

Primary Objectives:

-To evaluate the clinical efficacy of enzalutamide in patients with high-risk prostate cancer with regards to: Time to disease progression defined by biochemical recurrence (BCR)

Secondary Objectives:

-To further evaluate the safety of enzalutamide in patients with high-risk prostate cancer

Patients will receive daily oral therapy with enzalutamide at 160mg (4 capsules) orally once daily (QD). Patients will continue on study until progressive disease, drug intolerability, consent withdrawal or completion of study at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically confirmed adenocarcinoma of the prostate.
* Patients must have undergone a Radical Prostatectomy (any surgical technique is permitted) within 3 months from study entry and have high-risk disease define by any of the following:

  * Pathological stage T3a, T3b, T4 (any grade or iPSA)
  * Gleason' sum ≥ 8 (any stage or iPSA)
  * Initial Pre-operative PSA ≥ 20ng/mL (any GS or pT stage)
  * Any stage/PSA/Gleason patients with a 35% or greater chance of biochemical failure at 5 years based on Kattan's nomogram http://nomograms.mskcc.org/Prostate/PostRadicalProstatectomy.
  * Patients with Lymph node (LN) positive disease, regardless of iPSA, pT stage or GS provided their post-operative PSA 6-8 weeks after surgery is ≤ 0.4ng/mL. (Lymph node dissection is desired but not mandated)
* Able to swallow the study drug and comply with study requirements.
* Patients must have normal organ and marrow function as defined below:

  * Testosterone ≥ 50 ng/dL per laboratory reference range
  * Baseline Post-RP PSA ≤ 0.4
  * Hemoglobin ≥ 10.0 g/dL independent of transfusion
  * Absolute neutrophil count ≥1,500/mcL
  * Platelet count ≥100,000/ìL
  * Serum albumin ≥ 3.5 g/dL
  * Serum potassium ≥ 3.5 mmol/L
  * Liver function: serum bilirubin < 1.5 x ULN (except for patients with documented Gilbert's disease) and AST or ALT < 2.5 x ULN

Exclusion Criteria:

* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment
* Prior radiotherapy to the prostate or pelvis (related to prostate cancer). Concurrent adjuvant radiation therapy is permitted once patient has been enrolled on trial.
* Prior use of Abiraterone acetate or cytotoxic chemotherapy for prostate cancer
* Prior androgen deprivation with Luteinizing hormone-releasing hormone (LHRH) is permitted provided that testosterone levels prior to study entry have recovered to normal limits per reference laboratory.
* No prior anti-androgen therapy (bicalutamide, flutamide or Nilutamide) is permitted
* Prior use of 5-alpha reductase inhibitors is permitted provided such medications were stopped 7-14 days prior to enrollment
* Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within 2 weeks of enrollment
* Active unresolved infection
* Known history of central nervous system (CNS) metastases
* Patients must have no known history of HIV
* Evidence of metastatic disease as evidenced by a CT or MRI of abdomen and pelvis and/or whole body bone scan (WBS). To be done prior to treatment start and up to 4 months prior to radical prostatectomy date.
* History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke, significant brain trauma). Also, history of loss of consciousness or transient ischemic attack within 12 months of enrollment.
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months prior to Screening;
  * Uncontrolled angina within 3 months prior to Screening;
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram (ECHO) or multi-gated acquisition scan (MUGA) performed within 3 months results in a left ventricular ejection fraction that is ≥ 45%
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  * Hypotension as indicated by systolic blood pressure < 86 mmHg at the Screening visit
  * Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG
  * Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening visit
* Gastrointestinal disorder affecting absorption (e.g., Gastrectomy, active peptic ulcer disease within last 3 months)
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.
* The effects of enzalutamide on the developing human fetus at the recommended therapeutic doses are unknown. Thus, men must agree to use adequate contraception (barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 6 months after the usage of enzalutamide. Should the patient's partner become pregnant or suspect she is pregnant while the patient is participating in this study, the patient should inform his treating physician immediately.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enzalutamide
Started | 42
Completed | 37
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Financial Concerns | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Clinical Efficacy of Enzalutamide
Description: Clinical efficacy is measured as time to disease progression defined by biochemical recurrence (BCR). BCR was defined as PSA ≥0.2ng/mL on 2 consecutive lab results or any PSA rise that resulted in subsequent therapy.
Time Frame: 2 years
Population: All participants who received treatment and had biochemical recurrence.
Measure: Median (Full Range); unit: months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 5
months | 31 [13 to 40]

2. Secondary Outcome: Safety of Enzalutamide
Description: The number of patients that experience adverse events related to the study drug. NCI Cancer Clinical Trials Common Toxicity Criteria (version 4.0) will be utilized.
Time Frame: 2 years
Population: All participants that received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 42
Participants | 41

3. Other Pre Specified Outcome: Impact of Enzalutamide on Circulating Tumor Cells (CTCs)
Description: Quantify mRNA levels of Survivin in CTCs obtained from patients pre- and post-treatment with enzalutamide using the Veridex Cell Search Profile kit.
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected while participants were on treatment up to 2 years (24 cycles).
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 2/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=42)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=42)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15)
Anemia (Blood and lymphatic system disorders) | 9 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (18)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Blood bilirubin increased (Investigations) | 2 (3)
Breast pain (Reproductive system and breast disorders) | 16 (18)
Cognitive disturbance (Nervous system disorders) | 4 (4)
Concentration impairment (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 11 (14)
Dizziness (Nervous system disorders) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 37 (49)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Gynecomastia (Reproductive system and breast disorders) | 31 (33)
Headache (Nervous system disorders) | 7 (10)
Hot flashes (Vascular disorders) | 10 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (18)
Hypertension (Vascular disorders) | 4 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (10)
Lymphocyte count decreased (Investigations) | 9 (15)
Memory impairment (Nervous system disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Nausea (Gastrointestinal disorders) | 8 (14)
Nervous system disorders - Other, specify (Nervous system disorders) | 7 (11)
Pain (General disorders) | 27 (37)
Paresthesia (Nervous system disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rhinitis infective (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Weight gain (Investigations) | 20 (30)
Weight loss (Investigations) | 11 (13)
White blood cell decreased (Investigations) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT01927627/Prot_SAP_000.pdf